CLINICAL TRIAL: NCT00690209
Title: Efficacy of Surgical Coronary Revascularization Associated With Stem Cells Injection in Patients With Severe Chronic Ischemic Heart Disease With Residual Viability. A Prospective, Controlled Pilot Trial.
Brief Title: By Pass Surgery With Stem Cell Therapy in Chronic Ischemic Cardiopathy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: CHU-0034
Record Dates: First submitted 2008-05-30; First posted 2008-06-04 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Ischemic Heart Disease
Keywords: Chronic ischemic cardiomyopathy with residual viability; surgical coronary revascularization; stem cell therapy; Chronic ischemic heart disease; severe impairment of global contractility left ventricular dilation; residual viability
MeSH Terms: conditions — Myocardial Ischemia

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Procedure: Autologous bone marrow derived stem cells myocardial transplantation

SUMMARY:
Surgical revascularization has proven its efficacy in term of morbidity and mortality in patients with multivessel coronary disease and poor left ventricular function. Nevertheless, if left ventricle is severely dilated, the improvement of global contractility and reduction of volumes is frequently absent after CABG even if substantial amount of myocardial viability is present. A value of > 140 ml for end systolic volume has been proposed as the cut off for the absence of recovery after revascularization.

Recently, a reduction of cardiac volumes and improvement of regional and global contractility has been demonstrated in patients with advanced ischemic heart disease, severe dilation of left ventricle and poor candidates for revascularization after injection of stem cells in territories with residual viability.

DETAILED DESCRIPTION:
The screening of patients will be performed after contrast coronar ventriculography realized for diagnostic or prognostic purpose.

Subsequently all patients will be evaluated by cardiac ce-MR and PET imaging for verification of inclusion criteria.

Patients will be allocated in a single blind manner to one of two therapeutic arms: surgical revascularization alone or surgical revascularization associated with autologous bone marrow derived stem cells injection in viable territories.

During the follow up evolution of left ventricular volumes and contractility will be analyzed by ce-MR and PET imaging at 1 year. Additionally patients' functional status will be assessed by metabolic stress tests and quality of life questionnaire at 6 months, 1 year and 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Chronic ischemic heart disease
* Left ventricular dilation (end systolic volume >140 ml)
* Poor global contractile function (ejection fraction <40%)
* Substantial amount of residual viability (>30% of left ventricle)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2008-05; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Evolution of left ventricular volumes and contractility Evolution of left ventricular volumes and contractility

SECONDARY OUTCOMES:
Functional status

CONTACTS AND LOCATIONS:
Overall Officials: Janusz Lipiecki, Dr, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- Departements of CardiacSurgery, Cardiology and Radiology, Clermont-Ferrand, France